CLINICAL TRIAL: NCT03949868
Title: Mindful Attention to Variability in Everyday Memory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Karyn Gunnet-Shoval, Sub-Investigator, Harvard University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB18-0247
Record Dates: First submitted 2019-05-13; First posted 2019-05-14 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Memory Lapse
Keywords: mindfulness; forgetfulness; Langerian mindfulness
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not aware of how the conditions differ, nor are they aware of how many conditions there are.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Mindfulness (Experimental): All participants in this condition will complete all measures online and over the phone at two points in time, including one narrative response at T1. They will also be instructed to complete a mindfulness intervention at home and respond to diary-type text messaging questions (all including questions about memory performance) twice daily for six days.
  Interventions: Behavioral: High Mindfulness
- Low Mindfulness (Experimental): All participants in this condition will complete all measures online and over the phone at two points in time, including one narrative response at T1. They will also be instructed to respond to diary-type text messaging questions (some related to memory performance) twice daily for six days.
  Interventions: Behavioral: Low Mindfulness
- Active control (Active Comparator): All participants in this condition will complete all measures online and over the phone at two points in time, including one narrative response at T1. They will also be instructed to respond to diary-type text messaging questions (none about memory performance) twice daily for six days.
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: High Mindfulness — Those in the "high mindfulness" group will also receive questions about their memory performance over the past 30 minutes in both the morning and evening for six days. In order to emphasize the variability in pain, participants will receive these text messages on a variable schedule. In addition, they will sent instructions every morning to pay attention to variability in their memory performance throughout the day and asked to report on how their memory performance is changing over time as a part of each text message prompt.
  Arms: High Mindfulness
Behavioral: Low Mindfulness — Those in the "low mindfulness" group, who will receive receive two text messages per day (one at at 9am and one at 8pm) for six days, each prompting them to write about the activity they are currently engaged in. They will also be prompted with the 9am text to report on their memory performance over the past 30 minutes.
  Arms: Low Mindfulness
Behavioral: Active control — Participants in the "active control" group will receive 2 text messages per day for six days (one at 9am and one at 8pm) asking them to report on the activity they are currently engaged in.
  Arms: Active control

SUMMARY:
Forgetfulness is a common complaint among middle and older adults, with the vast majority of these complaints not rooted in established causes or diagnoses. The contents of these subjective cognitive complaints (SCC) include difficulty retrieving specific words (e.g., names of people or places), misplacing common items (e.g., keys or eyeglasses), and prospective memory failures (e.g., forgetting appointments and reasons for entering a room). One study found that 54% of people in a sample composed of 15,000 adults over the age of 55 reported that they had some difficulty remembering things over the past year. In the subsample composed of individuals aged 85+, this figure increased to 62%.

While some experiences of forgetting can be partially explained by age-related cognitive decline, problems with retrieval processes can be attributed to a host of other factors including stress and anxiety, lack of sleep, and side effects from medications. Even with all of these other possible aspects at play, older adults tend to attribute everyday instances of forgetting to uncontrollable factors including age. Moreover, while society tends to associate forgetting with the elderly population, young adults also report the experience of forgetting. There is reason to suspect that while older adults tend to experience more instances of forgetting than they did as younger adults, they also pay more attention to instances of forgetting, gathering evidence that they are declining. Every instance of forgetting can confirm that one is in the midst of decline. This process is a type of confirmation bias: Every time an older adult notices an instance of forgetting, he/she confirms that the self fits within the larger negative age stereotype. The present study investigates the Attention to Variability Paradigm. Specifically the participants will pay attention to how memory performance fluctuates throughout the day. Primary outcomes will be memory efficacy beliefs and memory performance on a telephone task.

DETAILED DESCRIPTION:
In the present study, the participants will be assigned to one of three groups: an active control group, a group asked to attend to everyday memory performance, and a group asked to notice variability in their everyday memory performance. The researchers hypothesize that the experimental groups will improve on memory outcomes more than those in the control group as a result of participation. The researchers hypothesize that when older adults are trained over 6 days to notice variability in memory ability the participants will report having more control over memory abilities then will the participants in the other two groups. The researchers also expect that the participants will show more improvement on a memory task than the participants in the other groups.

The researchers will take measurements of memory efficacy beliefs and memory performance at 2 timepoints (T0=baseline, T1= immediately after the 6 days of text messages). All surveys will be collected online via the Qualtrics.com platform.

ELIGIBILITY:
Inclusion Criteria:

* Age: 65-80
* An expressed concern or anxiety about memory performance (Responding "YES" when asked if concerned about memory at all)
* Fluent in English
* Owns a smartphone

Exclusion criteria:

* The presence of cognitive impairment (more than 2 incorrect responses) on the Short Portable Mental Status Questionnaire (SPMSQ), an instrument developed to assess cognitive functioning over the phone.
* The presence of any medical conditions that affect cognitive ability, such as stroke, acquired brain injury, dementia, and other neurological disorders or illnesses, or untreated hypertension.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Everyday Memory Questionnaire-Revised (EMQ-R; Royle & Lincoln, 2008) | 2 minutes
  This 13-item self-report scale measures subjective memory failures. Namely, respondents are asked to indicate whether or not they had experienced certain memory failures within the past 24 hours (e.g., "Did you find that a word was "on the tip of your tongue" - you knew what it was but could not quite find it?). Following the 13 yes/no questions about one's memory functioning, participants are asked to rate how stressful these failures are on a scale of 0-10 with 0 indicating "not at all stressful" to 10 indicating "very stressful." The final question asks the participant to compare their memory functioning that day compared to other days ("much worse than usual, a little worse than usual, same as usual, somewhat better than usual, much better than usual"). This 13-item version was shortened from the original 28-item version (Sunderland, Watts, Baddeley, & Harris, 1986).
Memory Controllability Inventory (MCI; Lachman, Bandura, Weaver, & Elliott, 1995) | 3 minutes
  The Memory Controllability Inventory is a 19-item Likert scale with questions about one's memory. Participants rate each statement from 1 (strongly disagree) to 7 (strongly agree). The MCI includes six subscales, including: Present Ability (e.g., "I can remember the things I need to."), Potential Improvement (e.g., "I can find ways to improve my memory"), Effort Utility (e.g., "If I work at it, I can improve my memory."), Inevitable Decrement (e.g., "There's not much I can do to keep my memory from going downhill.", Independence (e.g., "As I get older I won't have to rely on others to remember things for me.", and Alzheimer's Likelihood (e.g., I think there's a good chance I will get Alzheimer's disease"). On all the subscales except Alzheimer's Likelihood, higher scores indicate higher levels of perceived personal control over one's memory.
Multifactorial Memory Questionnaire (MMQ; Troyer & Rich, 2002). | 3 minutes
  The Multifactorial Memory Questionnaire is a 54-item self-report scale, which asks about overall satisfaction with one's memory ("MMQ-Contentment"), one's perceived memory ability ("MMQ-Ability"), and the extent to which one employs memory strategies ("MMQ-Strategy"). The MMQ-Contentment asks respondents to rate each item on a scale of 1 (strongly agree) to 5 (strongly disagree), with 3 indicating "undecided." An example of the "Contentment" subscale is "I am generally pleased with my memory ability." The MMQ-Ability subscale asks respondents to rate 20 different memory mistakes on a scale of 1 (all the time) to 5 (never). An example of the "Ability" subscale is "Forgot an appointment." The MMQ-Strategy subscale asks respondents to rate how often they used a given memory strategy on a scale of 1 (all the time) to 5 (never). An example of a strategy included in this subscale is, "Use a timer or alarm to remind you when to do something."
Brief Test of Adult Cognition by Telephone with Stop-and-Go Switch Task (BTACT; (Tun & Lachman, 2006) | 20 minutes
  The BTACT is a neuropsychological battery based off well-known laboratory tasks and modified versions of well-established psychometric tests. The BTACT, which is proctored over the phone, is designed to be sensitive to performance a range of cognitive abilities in older adults without cognitive impairments including: episodic verbal memory (both immediate and delayed list recall of 15 unrelated words of the Rey Auditory-Verbal Learning Test, Rey, 1964), working memory span (backwards digit span, Wechsler, 1997) and language verbal fluency. We also included the optional Stop-and-Go switch task to test task-switching ability/inhibitory control. Two versions of the test (Form A and Form B) are available for repeated measurement. This test has demonstrated good construct validity and test-retest reliability (Lachman, Agrigoroaei, Tun, & Weaver, 2014). Moreover, the assessment's authors found no difference in performance between individuals who took the test over the phone vs. in person.

SECONDARY OUTCOMES:
Langer Mindfulness Scale (LMS-14; Pirson, Langer, Bodner, & Zilcha, 2012) | 2 minutes
  Trait mindfulness is assessed using the Langer Mindfulness Scale (LMS-14), a 14-item Likert scale (1= Strongly disagree to 7 = Strongly agree) which includes three factors: novelty seeking, novelty producing, and engagement. The authors reported good psychometric properties.
Positive and Negative Affect Schedule (PANAS; Watson, Clark, & Tellegen, 1988) | 2 minutes
  The Positive and Negative Affect Schedule prompts participants to consider twenty mood states and rate each one a scale of 1 to 5 with 1 indicating "very slightly or not at all" and 5 indicating "extremely". Specifically, we used the variation of the scale that asks participants to rate their current mood (i.e., "the way you feel now, that is, at the present moment", Watson et al., 1988, pg. 106). PANAS has been shown to include two factors, namely, positive affect (PA) and negative affect (NA). The two factors are calculated by summing the 10 positive emotions and the 10 negative emotions. The PANAS referring to mood states in the present moment has excellent internal consistency with the PA alpha coefficient = .89 and the NA alpha coefficient = .85.
Image of Aging Scale (Levy, Kasl, & Gill, 2004). | 2 minutes
  This scale prompts participants to rate 18 characteristics on how well they describe "old people in general." Participants rate the extent to which each characteristic matches one's image of aging using a 7-point Likert scale with 0 indicating "does not match my image" to 6 indicating that the characteristic "completely matches my image". In the development of this scale, eighteen traits were conceptually matched across nine dimensions so that positive and negative age-based stereotypes each had an opposite (e.g., "walks slowly" and "active"). These nine domains included activity, appearance, cognition, death, dependence, personality, physical health, social relationships, and will to live. The Image of Aging Scale has good psychometric properties.
Subjective Age Measure (Barak & Schiffman, 1981). | 2 minutes
  Subjective age was assessed with Barak and Schiffman's subjective age measure (1981), which taps into cognitive, psychological, biological, and social domains of the subjective age construct. Specifically, the measure prompts participants to report on "feel age" (i.e., how old participants feel), "look age" (i.e., how old participants believe they look), "do age" (i.e., how old participants believe they act), and "interest age" (i.e., the age group they believe would share their interests). Specifically, we calculated the difference between their actual age and subjective age. The authors reported good internal consistency and reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States